CLINICAL TRIAL: NCT04774146
Title: Quantification of Silicone Oil Emulsification After Pars Plana Vitrectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Sponsor
Other Study IDs: 1/2000
Record Dates: First submitted 2020-09-16; First posted 2021-03-01 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-09

CONDITIONS: PArs Plana Vitrectomy; Retinal Detachment; Silicone Oil Droplets on Intraocular Lens
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — lavage fluid (Balanced Salt Solution) irrigating the vitreous chamber
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- triple air fluid exchange: those undergoing triple air fluid exchange
  Interventions: Procedure: pars plana vitrectomy
- irrigation: those undergoing vitreous chamber irrigation with comparable volume of BSS
  Interventions: Procedure: pars plana vitrectomy

INTERVENTIONS:
Procedure: pars plana vitrectomy — silicone oil active aspiration and isovolumetric BSS replacement followed by irrigation and /o gas fluid exchange

SUMMARY:
silicone oil tamponade removal after previous injection of complicated retinal detachment can be achieved with active suction followed by triple air-fluid exchange or prolonged lavage of the vitreous chamber to remove emulsification. Purpose of the study is to compare the amount of silicone oil emulsification droplets within the lavage fluid in case of air exchange and simple lavage to compare which technique removed the highest percentage of emulsion. This is achieved by comparing consecutive samples of lavage fluid

DETAILED DESCRIPTION:
silicone oil tamponade removal after previous injection of complicated retinal detachment can be achieved with active suction followed by triple air-fluid exchange or prolonged lavage of the vitreous chamber to remove emulsification. Purpose of the study is to compare the amount of silicone oil emulsification droplets within the lavage fluid in case of air exchange and simple lavage to compare which technique removed the highest percentage of emulsion. This is achieved by comparing consecutive samples of lavage fluid.

Therefore consecutive patients scheduled to SiO removal with triple air exchange or vitreous chamber lavage are enrolled and 3 samples of intraocular fluid aspirated during the fluid exchange procedure sent to the lab for SiO emulsion count and quantification.

ELIGIBILITY:
Inclusion Criteria:

* previous silicone oil tamponade after pars plana vitrectomy
* age >18 years
* Attached retina

Exclusion Criteria:

* unwilling or unable to participate,
* previous multiple eye surgery
* History of Trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing previous retinal detachment surgery with pars plana vitrectomy with silicone oil tamponade
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-11-03 (Estimated)

PRIMARY OUTCOMES:
number of silicone oil emulsification droplets per volume unit | 6 months after primary surgery
  number of silicone oil emulsification droplets per volume unit. Fluid taken from the vitreous chamber during surgery is subsequently analyzed. Therefore time frame is just one: after taking all samples they are analyzed to count oil droplets per volume unit

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Rossi, Study Director — IRCCS Policlinico San MArtino
Locations (1):
- IRCCS Policlinico San Martino, Genova, RM, Italy

IPD SHARING:
Plan to Share IPD: No